CLINICAL TRIAL: NCT03549312
Title: Evaluation of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) Switch Followed by Sofosbuvir/Velpatasvir (SOF/VEL) Antiviral HCV Therapy Followed by Bictegravir/Emtricitabine/Tenofovir Alafenamide (B/F/TAF) Simplification in HIV-HCV Co-Infected Subjects on Opioid Substitution Therapy - A Pilot Feasibility Study
Brief Title: Switch to Genvoya Followed by HCV Therapy With Epclusa Followed by Simplification of HIV Therapy With Biktarvy in Patients With HIV-HCV Co-Infected Subjects on Opioid Substitution Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Alexander Wong, MD, Assistant Professor, Division of Infectious Diseases, Saskatchewan Health Authority - Regina Area
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB-17-22
Record Dates: First submitted 2018-04-22; First posted 2018-06-08 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: HIV-1-infection; Hepatitis C, Chronic; Methadone Dependence; Opioid Dependence; Bone Diseases, Metabolic; HIV/AIDS; Co-infection; Buprenorphine Dependence; HCV Coinfection
Keywords: HIV; Hepatitis C; Methadone; HIV/HCV Co-Infection; Opioid Substitution Therapy; Buprenorphine/Naloxone
MeSH Terms: conditions — Hepatitis C, Chronic; Opioid-Related Disorders; Bone Diseases, Metabolic; Acquired Immunodeficiency Syndrome; Coinfection; Hepatitis C | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; elvitegravir; sofosbuvir-velpatasvir drug combination; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Switch to Genvoya Followed By HCV Therapy Then Start Biktarvy (Experimental): Oral Genvoya 150/150/200/10 mg & Epclusa 400/100 mg once daily. Once completed HCV therapy, switch anti-retroviral treatment to Oral Biktarvy 50/200/25 mg.
  Interventions: Drug: Genvoya; Drug: Epclusa; Drug: Biktarvy

INTERVENTIONS:
Drug: Genvoya — Switching to Genvoya for 48 weeks in patients with HIV/HCV co-infection and stably suppressed HIV RNA, prior to starting HCV treatment, while receiving methadone or buprenorphine/naloxone as opioid substitution therapy.
  Plasma HIV-1 RNA < 50 copies/mL at weeks 4, 12, 24, 36 and 48.
  Other Names: Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide
Drug: Epclusa — HCV therapy with direct-acting-antiviral therapy with Epclusa in HIV-HCV co-infected patients with suppressed HIV RNA, receiving methadone as opioid substitution therapy.
  Plasma HCV RNA viral load at weeks 12, 24, 36, 48, 72 and 96.
  Other Names: Sofosbuvir and Velpatasvir
Drug: Biktarvy — Switching to Biktarvy for 48 weeks in patients with HIV previously treated with Genvoya, stably supressed HIV RNA, while receiving methadone or buprenorphine/naloxone as opioid substitution therapy.
  Plasma HIV-1 RNA < 50 copies/mL at weeks 52, 60, 72, 84 and 96.
  Other Names: Bictegravir, Emtricitabine and Tenofovir Alafenamide

SUMMARY:
The study hypothesis is to determine the feasibility of switching HIV-HCV co-infected patients receiving methadone or buprenorphine/naloxone as opioid substitution therapy with suppressed HIV RNA viral load on current antiretroviral therapy to elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF, Genvoya™) followed by 12 weeks of HCV antiviral therapy with sofosbuvir/velpatasvir (SOF/VEL, Epclusa™), followed then by switch to bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF, Biktarvy™) for an additional 48 weeks.

DETAILED DESCRIPTION:
This clinical study is a phase IV, prospective, open-label study that is being conducted in 25 participants over the age of 18 on stable antiretroviral therapy with documented HIV viral suppression who have received opioid substitution therapy (OST) for at least three months. The study is designed to assess the feasibility of the switch from a participant's current antiretroviral therapy (ART) regimen to Genvoya, followed shortly thereafter by initiation of Epclusa for treatment of HCV co-infection with subsequent optimization of the ART regimen to Biktarvy in patients co-infected with HIV and HCV receiving methadone or buprenorphine/naloxone as OST. Participants will be recruited from the Infectious Diseases Clinic (IDC) in Regina, a tertiary referral site that cares for a large number of patients living with HIV and viral hepatitis.

Eligible participants will have baseline investigations performed, including measures of renal parameters and bone mineral densitometry, and will be switched from their current antiretroviral regimen to Genvoya for the first 12 weeks of the study. Various reasons for switching may play a role in clinician decision-making, including simplification, improved tolerability, an improved metabolic risk profile, etc. The primary drawbacks to Genvoya in clinical practice include the potential for drug-drug interactions due to the presence of cobicistat, and the relatively low so-called "genetic barrier" of resistance, meaning that sub-optimal adherence may be more likely to result in antiretroviral resistance. Participants must already be fully suppressed at the time of screening to be enrolled in the study, as well as having been stable on OST for at least three months, in order to reduce the risk of poor adherence.

After the switch to Genvoya occurs, participants will be seen at weeks 1 and 4 to assess for adverse events, including any changes in OST dosing. Laboratory testing will be performed as per standard of care with CD4 counts and HIV viral loads checked at weeks 4 and 12 to ensure stable virologic suppression following switch of ART. After 12 weeks of Genvoya, provided that participants remain stably suppressed in terms of their HIV, they will then receive 12 weeks of Epclusa to treat their chronic HCV infection while continuing to take Genvoya. Participants are allowed to have any HCV genotype and may have stage 0-4 liver fibrosis as assessed by transient elastography, but may not have decompensated cirrhosis or hepatocellular carcinoma. Participants will be followed at weeks 13, 16 and 24 with clinical assessments performed, and repeat HCV viral loads at weeks 16 and 24 (end of HCV treatment) as per standard of care. Participants will be seen at weeks 36 and 48 and have their HCV viral loads performed to determine whether they have achieved a sustained virologic response 12 and 24 weeks following end of HCV therapy, which defines HCV cure. Bone mineral densitometry will be performed at week 48 to determine any interval change in bone mineral density has occurred between study initiation and week 48.

After the 48 weeks of treatment with Genvoya, participants who agree will be switched to a modern unboosted ARV regimen consisting of Biktarvy through a 48 week extension phase. Biktarvy is approved by Health Canada as an unboosted integrase-inhibitor based single-tablet regimen with once-daily dosing and a small pill size, which facilitates adherence to treatment. Due to the presence of bictegravir, Biktarvy is likely to have a higher "genetic barrier" of resistance than Genvoya, and the lack of boosting significantly decreases the risk of drug-drug interactions. During the extension phase, participants will be seen at weeks 49, 52, 60, 72. 84 and 96 for clinical assessments with HIV viral loads, CD4 counts and standard of care laboratory testing. Bone mineral densitometry will be performed at week 96 to determine any interval change in bone mineral density has occurred between study initiation and week 96.

At each visit, participants will see a study coordinator and have vital signs performed, a review of their concurrent medications including any changes in their methadone dosing, review for any adverse events, and weight and height measurements. Laboratory investigations and urine drug screens will be performed as per current standards of care. Validated questionnaires assessing whether the participant is having any symptoms or signs of opioid withdrawal or overdose as well as determining treatment satisfaction with their new antiretroviral regimen. will be administered at each visit. Each visit is anticipated to take approximately 60-90 minutes, and the appointment for bone mineral density testing will take no longer than 2 hours to complete with waiting time included. All study medication will be provided during study period but not after study completion.

At study conclusion, demographic and other baseline variables will be summarized using percentage, mean, median, standard deviation and interquartile range as appropriate. The proportion of subjects achieving the various endpoints and the associated 95% confident interval will be calculated. Adverse events will be summarized by grade and relationship to treatment in addition to presenting the data in a listing format.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Females, 18 years or older
2. HIV infected (ELISA with western blot confirmation)
3. HCV RNA positive for minimum of 6 months / Genotype 1-6
4. Prescribed a combination ART regimen (cART) that may include any DHHS recommended or alternative regimens, which the treating physician considers is appropriate for their patient, except E/C/F/TAF or B/F/TAF at any point previously.
5. HIV RNA ≤ 50 c/mL at screening and ≤ 200 c/mL for at least 3 months prior to screening.
6. CD4 ≥ 200 cells/uL at screening.
7. Stage 0 to 4 fibrosis.
8. On methadone or buprenorphine/naloxone as OST for at least 3 months prior to screening and deemed stable on OST by the investigator.
9. Treatment naïve to all anti-HCV therapy, or treatment experienced but with no previous exposure to NS5A inhibitors.
10. Ability to remain adherent to medications and study protocol as per investigator opinion
11. Must be willing and able to understand the requirements of study participation and provide signed and dated written informed consent prior to screening.
12. Female subjects are willing to use acceptable methods of birth control as defined in the protocol.

Exclusion Criteria:

1. Have received any anti-HCV therapy previously with NS5A inhibitors. Previous treatment regimens allowed may include pegylated interferon, ribavirin, 1st generation NS3/NS4 protease inhibitors (telaprevir or boceprevir), and sofosbuvir.
2. Have any evidence of decompensated liver disease including ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy, or other symptoms suggestive of advanced liver disease. For cirrhotic patients with Child-Pugh Class B or C or with Pugh-Turcotte (CPT) score greater than 6 must be excluded.
3. Co-infection with hepatitis B.
4. Has cirrhosis and liver imaging within 6 months of Day 1 showing evidence of hepatocellular carcinoma (HCC), or is under evaluation for HCC.
5. Concomitant use of drugs with contraindication or drug-interactions with E/C/F/TAF on Day 1 visit or B/F/TAF on Week 48/0E visit. However, the use of any concomitant drugs with contraindication with SOF/VEL are to be stopped during the weeks of treatment (i.e. week 12-24), and only after the Principal Investigator's permission, may the use of these drugs may be continued or restarted after week 24 visit (i.e. end of SOF/VEL therapy).
6. Have any active contraindication to the use of methadone, as listed in the product monograph for methadone and listed below, unless deemed acceptable based on the Principal Investigator's judgement:

   1. Patients who are hypersensitive to the active substance (methadone hydrochloride) or other opioid analgesics or to any ingredient in the formulation.
   2. Patients with a known or suspected mechanical gastrointestinal obstruction.
   3. Patients with a suspected surgical abdomen.
   4. Patients with acute asthma or other obstructive airway, and status asthmaticus.
   5. Patients with acute respiratory depression, elevated carbon dioxide levels in the blood, and corpulmonale.
   6. Patients with acute alcoholism, delirium tremors, and convulsive disorders.
   7. Patients with severe central nervous system depression, increased cerebrospinal or intracranial pressure, and head injury.
   8. Patients taking monoamine oxidase (MAO) inhibitors (or within 14 days of such therapy).
   9. Patients with diarrhea associated with pseudomembranous colitis caused by cephalosporins, lincomycins (including topical clindamycin) or penicillin, or to patients having diarrhea caused by poisoning, until toxic material has been eliminated from the gastrointestinal tract.
7. Concomitant use of alcohol to a degree deemed by the investigator to be dangerous in conjunction with administration of methadone.
8. Has documented historic resistance to any of the components of E/C/F/TAF or B/F/TAF.
9. Has an eGFR (by MDRD equation) < 30 mL/min/1.73m2.
10. Is pregnant, breast-feeding, or planning or suspected to get pregnant.
11. Has any reason, in the opinion of the investigator, which would make the candidate inappropriate for participation in an investigative study involving oral medications.
12. Involved in any other interventional HIV or HCV study during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-07-21 (Estimated); Study Completion 2021-06-22 (Estimated)

PRIMARY OUTCOMES:
Feasibility assessment: participants approached, screened and enrolled in the study along with completed study visits | Up to 48 weeks on Genvoya and 12 weeks of Epclusa and 48 weeks of Biktarvy
  Feasibility will be measured by collecting data on the number of participants approached, screened and enrolled. In addition, feasibility will be assessed by proportion of completed study visits as outlined in the protocol.
Assessment of incidence of screen failures | Week 96
  Screen failures will be assessed by drug-drug interactions, prior documented resistance to any component of Genvoya or Biktarvy, non-adherence to opioid substitution therapy or antiretroviral therapy.
Adherence | Week 96
  Adherence will be assessed at key time points of the study and will be determined by patient self-report and pill count at each study visit and by reviewing the accountability logs provided to the pharmacists to keep track of dispensed and returned pills or bottles for subjects receiving their study medication from their pharmacy with their OST.

SECONDARY OUTCOMES:
HCV clearance post Epclusa therapy | Weeks 24 and 48
  Proportion of participants with HCV RNA <12 copies/mL (c/mL) at Week 24 and Week 48
Sustained HIV Viral Load Suppression | Weeks 4, 12, 24, 36, 48, 52, 60, 72, 84 and 96
  Proportion of participants who maintain suppressed HIV Viral Load (i.e. plasma HIV-1 RNA <= 50 copies/mL)
Discontinuation of study medication due to adverse events | 96 weeks
  Proportion of participants discontinuing study medications due to adverse events (overall and liver enzyme abnormalities
Adjustments to methadone or buprenorphine/naloxone dosing over study duration | 96 weeks
  Proportion of participants who required any changes in the methadone or buprenorphine/naloxone dosing deemed secondary to the use of Genvoya, Epclusa or Biktarvy
Opioid withdrawal or overdose symptoms over study duration | 96 weeks
  Proportion of participants who experience opioid withdrawal or overdose symptoms while receiving Genvoya, Epclusa or Biktarvy and methadone or buprenorphine/naloxone as OST through 96 weeks of study, as per standardized survey measures.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Wong, MD, Principal Investigator — Saskatchewan Health Authority - Regina Area
Locations (1):
- Saskatchewan Health Authority, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No